CLINICAL TRIAL: NCT05696340
Title: Access to Pediatric Rheumatology Centers for JIA Patients: Factors Associated With Time to Access Pediatric Rheumatology Centers
Acronym: AJILITT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Research on Healthcare Performance Lab U1290 (Other)
Responsible Party: Sponsor
Other Study IDs: 2022 CHAUSSET AJILITT
Record Dates: First submitted 2022-12-22; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-12

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: qualitative research; access to care; time to referral; health literacy
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- JIA patients: Children diagnosed with JIA between 4 and 24 months before the start of the study, treated and followed in a pediatric rheumatology center (old enough to answer the questions)
  Interventions: Other: semi-structured interview
- Parents of JIA patients: Parents of a child diagnosed with JIA between 4 and 24 months prior to the start of the study (treated and followed in a pediatric rheumatology center)
  Interventions: Other: semi-structured interview
- Health care professionals: Physician with experience in the initial management of JIA patients (between symptom onset and first visit with a pediatric rheumatologist)
  Interventions: Other: semi-structured interview

INTERVENTIONS:
Other: semi-structured interview — Subjects will be recruited in a purposive, non-randomized manner. Data will be collected to obtain a sufficient diversity of perspectives on the topic, while maintaining sufficient homogeneity for analysis.
  The number of participants cannot be determined in advance; it will be determined after data saturation.

SUMMARY:
JIA patients, their parents, and the health care professionals experience the complexity of the initial care pathway. The aim of the study is to explore the referral pathway to access pediatric rheumatology centers for JIA patients. The exploration will aim to identify the barriers and facilitators of referral, based on the conceptual framework of the health literacy. The investigators will conduct a qualitative study using semi-structured interviews. The perspectives of parents/children/health care professionals will be crossed to enrich the data.

ELIGIBILITY:
Inclusion Criteria:

Children:

* age > 11 years
* JIA diagnosed between 4 and 24 months prior to the start of the study

Parents:

- parent of a child with JIA diagnosed between 4 and 24 months prior to the start of the study

Health care professional:

* Physician with experience in the initial management of children with JIA (between symptom onset and first visit with a pediatric rheumatologist).

Exclusion Criteria:

For all participants:

* Refusal to participate in interviews
* Presenting a health condition incompatible with an interview
* Participants with inadequate French to take part in semi-structured interviews

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children, adolescents, their parents, and the health care professionnals who have experienced the initial care pathway for JIA (between symptom onset and first visit with a pediatric rheumatologist).
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Experience and views of barriers and solutions to the referral to pediatric rheumatology center for JIA patients | About 1 hour
  Through semi-structured interviews, the study will reconstruct the referral pathway to the pediatric rheumatology center for JIA patients.
  * For patients and their parents, the interviews will focus on their experiences of the health care system, their feelings about interactions with health professional, their expectations and the elements that led to the parents' decision regarding their child's health.
  * For health care professionals, the interviews will focus on their experience in managing children with JIA (from the symptom onset to the first visit with the pediatric rheumatologist), the difficulties they encountered, and the improvements to be made in training and communication.

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie CHAUSSET, Study Director — University Hospital, Clermont-Ferrand
Locations (4):
- France (4):
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Hospices Civils de Lyon, Lyon
  - APHP, Paris
  - Hopital Nord Franche-Comté, Trévenans

REFERENCES:
- [Background] Chausset A, Pereira B, Echaubard S, Merlin E, Freychet C. Access to paediatric rheumatology care in juvenile idiopathic arthritis: what do we know? A systematic review. Rheumatology (Oxford). 2020 Dec 1;59(12):3633-3644. doi: 10.1093/rheumatology/keaa438. PMID 32940701
- [Background] Davies K, Cleary G, Foster H, Hutchinson E, Baildam E; British Society of Paediatric and Adolescent Rheumatology. BSPAR Standards of Care for children and young people with juvenile idiopathic arthritis. Rheumatology (Oxford). 2010 Jul;49(7):1406-8. doi: 10.1093/rheumatology/kep460. Epub 2010 Feb 19. No abstract available. PMID 20173199
- [Background] Scott C, Chan M, Slamang W, Okong'o L, Petty R, Laxer RM, Katsicas MM, Fredrick F, Chipeta J, Faller G, Pileggi G, Saad-Magalhaes C, Wouters C, Foster HE, Kubchandani R, Ruperto N, Russo R. Juvenile arthritis management in less resourced countries (JAMLess): consensus recommendations from the Cradle of Humankind. Clin Rheumatol. 2019 Feb;38(2):563-575. doi: 10.1007/s10067-018-4304-y. Epub 2018 Sep 28. PMID 30267356
- [Derived] Chausset A, Freychet C, Lohse A, Belot A, Merlin E, Echaubard S, Schott AM, Lachal J. Diagnosis journey for children with juvenile idiopathic arthritis: a qualitative study. Arch Dis Child. 2024 Nov 19;109(12):1003-1009. doi: 10.1136/archdischild-2024-327426. PMID 39174297